CLINICAL TRIAL: NCT03898336
Title: Eat2beNICE Vitamins and Nutrients as Supplementation for Impulsivity, Irritability, and Compulsivity
Acronym: VANTASTIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Central Institute of Mental Health, Mannheim (Other); University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VANTASTIC STUDY
Record Dates: First submitted 2019-02-07; First posted 2019-04-01 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Impulsive Behavior
MeSH Terms: conditions — Impulsive Behavior

STUDY DESIGN:
Intervention Model Description: double-blind placebo controlled following open label phase
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- broad-spectrum micronutrients (Experimental): broad-spectrum micronutrients description: capsules containing a blend of Vitamin B3 (NADH), Vitamin B6 (pyridoxal-5-phosphate), folic acid (5-MTHF), Vitamin B12 (methylcobalamin), Vitamin D3 (25-hydroxyvitamin D3), Magnesium (magnesium oxide), Zinc (zinc methionine), Iron (ferric phosphate), Selenium (selenomethionine), Phospholipids, L-carnitine (L-carnitine-L-tartrate)
  Interventions: Other: broad-spectrum micronutrient
- placebo (Placebo Comparator): capsules containing placebo
  Interventions: Other: placebo

INTERVENTIONS:
Other: broad-spectrum micronutrient — daily intake of capsules containing a blend of Vitamin B3 (NADH), Vitamin B6 (pyridoxal-5-phosphate), folic acid (5-MTHF), Vitamin B12 (methylcobalamin), Vitamin D3 (25-hydroxyvitamin D3), Magnesium (magnesium oxide), Zinc (zinc methionine), Iron (ferric phosphate), Selenium (selenomethionine), Phospholipids, L-carnitine (L-carnitine-L-tartrate)
  Arms: broad-spectrum micronutrients
Other: placebo — daily intake of capsules
  Arms: placebo

SUMMARY:
Impulsivity, irritability and compulsivity are cross-disorder symptom domains, which affect a significant proportion of adolescents.

Predominately as part of attention deficit hyperactivity disorder (ADHD) but also as symptom domains without a diagnosis of ADHD, impulsivity and irritability cause serious burden. Furthermore, treatment options and their effects are limited.

Previous studies with different study designs assessing micronutrients for the treatment of impulsivity / ADHD in children and adults have reported positive benefits as well as a very good tolerability. However, more research is required; in particular controlled studies with adolescents, cross-disorder approaches and studies investigating long-term effects are missing.

The focus of this study is to investigate the effect of micronutrients on impulsivity, irritability and compulsivity in children and adolescents between 11 and 18 years of age with a high level of impulsivity and irritability with or without a diagnosis of attention deficit hyperactivity disorder (ADHD).

The investigators intend to include 210 children and adolescents (n=110 in Germany) with a high level of impulsivity and irritability.

The study is divided in two phases. An initial 10-week double blind, placebo-controlled treatment phase with broad-spectrum micronutrients is followed by a 10-week open-label treatment phase. The study assessments will be performed during five study visits and a follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 11;0 - 17; 6 years at initial inclusion
* Subjects with a high level of impulsivity/ irritability based on a CGI-S-score ≥ 4 and a parent-rated Affective Reactivity Index (ARI) score ≥ 5 indicating a high level of multi-dimensional irritability
* Subjects with or without a research diagnosis of attention deficit hyperactivity disorder (ADHD). ADHD has to be confirmed by structured diagnostic interview (ADHD section of Kiddie Schedule for Affective Disorders and Schizophrenia (K-SADS))
* Deemed reliable and compliant with the protocol (including the ingestion of as many capsules as prescribed by the investigator)
* Ability to comprehend and speak the native language of the country in which the assessments take place
* Signed informed consent by parents or legal representative
* Signed informed assent by child or adolescent (indicating that the subject is aware of the investigational nature and the core aspects of the study and the study is run in accordance with the ICH GCP guideline E6 (R2) (2016))

Exclusion Criteria:

* Subject is being treated with a medication that might, in the opinion of the investigator, pose a safety risk for the subject when participating in this study
* Intellectual disability (based on available IQ or the clinical opinion of the investigator, taking into account relevant psychosocial information, e.g. educational level)
* Any known abnormality of mineral metabolism (e.g., Wilson's disease, haemochromatosis)
* History of or present clinically relevant somatic or psychiatric acute or chronic disorder that, in the opinion of the investigator, might confound the results of tolerability/safety assessment, or prohibit the patients from completing the study, or would not be in the best interest of the patient.
* Subject has taken any kind of food supplement containing vitamins, minerals and/or trace elements within 30 days prior to entering the study
* Subject has unstable treatment conditions (current changes in medication and/or psychotherapy) that might in the opinion of the investigator confound the results of the study with respect to impulsivity/irritability.
* Subject has a documented allergy, hypersensitivity, or intolerance to any of the ingredients of the investigational product
* Subject has taken another investigational product or taken part in a clinical study within 30 days prior to entering the study

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 210 (Estimated)
Dates: Start 2019-09-18 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
response rate at end of placebo-controlled phase defined as CGI-I score with focus on impulsivity of 1 or 2 [=very much improved or much improved] plus reduction in Affective Reactivity Index (ARI) total score of at least 30% compared to baseline | 10 weeks (end of placebo-controlled phase)
  The primary objective is to investigate the double-blind placebo controlled (10 weeks) effects of broad-spectrum micronutrients in highly impulsive children and adolescents (10-18 years; N=180 in total) with a high level of impulsivity with or without diagnosis of attention deficit hyperactivity disorder (ADHD). The primary outcome measure is the response rate at the end of the placebo-controlled phase. Response is defined as a Clinical Global Impression - Improvement score (CGI-I, Guy 1976; NIMH 1985) with a focus on impulsivity of 1 or 2 [=very much improved or much improved] plus a reduction in the Affective Reactivity Index (ARI, parent-rated, Stringaris et al. 2012) total score of at least 30% compared to baseline.

SECONDARY OUTCOMES:
Change in Clinician rating of compulsivity | every 10 weeks over the whole study period of 20 weeks (10 weeks placebo-controlled phase followed by 10 weeks open label)
  Children´s Yale-Brown Obsessive-Compulsive Scale (CY-BOCS, Scahill et al., 1997)
Change in the rating of irritability | every 10 weeks over the whole study period of 20 weeks (10 weeks placebo-controlled phase followed by 10 weeks open label)
  Perceived Stress Scale (PSS-10, Taylor 2015)
Change in sleep problems | every 10 weeks over the whole study period of 20 weeks (10 weeks placebo-controlled phase followed by 10 weeks open label)
  Sleep problems (5-item questionnaire, self-rating of sleep problems)
change in motor activity (optional) | at baseline and after 10 weeks of study participation
  mHealth (movisens DataAnalyzer software)
Change in ADHD symptom severity total score | every 10 weeks over the whole study period of 20 weeks (10 weeks placebo-controlled phase followed by 10 weeks open label)
  Swanson, Nolan and Pelham Rating Scale (SNAP, Swanson et al. 2001)
change in rating of aggression | every 5 weeks over the whole study period of 20 weeks (10 weeks placebo-controlled phase followed by 10 weeks open label)
  Retrospective Modified Overt Aggression Scale (R-MOAS, Blader et al. 2010)
Rates of adverse events of the treatment groups in comparison to placebo group | every 5 weeks over the whole study period of 20 weeks (10 weeks placebo-controlled phase followed by 10 weeks open label)
  Compare rates of adverse events of the treatment groups to placebo group to assess safety and tolerability
change in treatment adherence | every 10 weeks over the whole study period of 20 weeks (10 weeks placebo-controlled phase followed by 10 weeks open label)
  assessed by Attitudes Towards Treatment questionnaire; total score 0-108; better Outcome: lower score

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Haege, Dr., Principal Investigator — Central Institute of Mental Health, Mannheim
Locations (1):
- Central Institute of Mental Health, Mannheim, Germany